CLINICAL TRIAL: NCT05993221
Title: Deconstructing Post Stroke Hemiparesis for Precision Neurorehabilitation
Brief Title: Deconstructing Post Stroke Hemiparesis
Acronym: TRACTs
Status: Recruiting | Type: Observational
Sponsor: Providence VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Lin, Neurologist, Core Investigator, Providence VA Medical Center
Other Study IDs: 1689966
Record Dates: First submitted 2023-07-06; First posted 2023-08-15 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
TRACTs (DeconsTructing Post StRoke HemipAresis for PreCision NeurorehabiliTation) is a single timepoint study that aims to deconstruct post-stroke deficits of the upper extremity into distinct components and relate these components to brain anatomy and physiology.

DETAILED DESCRIPTION:
Veterans will be recruited through the Providence Veterans Affairs Medical Center and will have research visits at the Providence VA Center for Neurorestoration and Neurotechnology (CfNN, centerforneuro.org). The research visits will span two to three days. The study will involve motor outcome measures, magnetic resonance imaging of the brain, and transcranial magnetic stimulation. The goal of this study is to associate post-stroke deficits of the upper extremity with brain anatomy and physiology.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a unilateral ischemic stroke occurring >6 months prior as documented in medical chart
* Upper extremity motor impairment as measured by Fugl-Meyer Upper Extremity Assessment ≤60
* Ability to follow simple instructions in English

Exclusion Criteria:

* Greater than moderate difficulty using the arm and hand pre-dating the stroke as assessed by the questions adapted from the QuickDASH outcome measure score on any question >= 3, which measures physical function and symptoms in people with difficulty using the arm and hand.
* Visual or auditory disorders resulting in the inability to see or hear, respectively, the stimuli presented as part of research sessions
* Inability to maintain a seated position for at least one hour
* Standard MRI exclusion (e.g., significant claustrophobia or inability to tolerate loud noises, cardiac pacemaker (unless MRI-safe), implanted device (deep brain stimulation) or metal in the brain, cervical spinal cord, or upper thoracic spinal cord)
* Standard (single-pulse) TMS exclusion which include (in addition to those listed for MRI) pregnancy/lactation/planning to become pregnant during the study, seizure disorder, and primary or secondary CNS tumors

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans who have sustained a unilateral ischemic stroke at least six months prior to recruitment with resulting upper extremity deficit(s).
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Arm Motor Assessment | Assessment occurs at one cross-sectional timepoint within 2 weeks of research consent
  This test provides information about the level of upper extremity motor impairment after stroke. It consists of a 33-item assessment, which provides a global assessment of upper extremity motor impairment. A rater observes 30 voluntary upper extremity motions, two tendon tap responses, and provides an ordinal rating (2 = near normal ability/response, 1 = partial ability, 0 = unable to perform/no response). The Fugl-Meyer Upper Extremity scale has excellent intra-rater reliability (0.99), inter-rater reliability (0.99), test-retest reliability (0.94-0.99), and internal consistency (0.97).

SECONDARY OUTCOMES:
Edinburgh Handedness Inventory | Assessment occurs at one cross-sectional timepoint within 2 weeks of research consent
  This screener is used to identify the handedness of participants prior to stroke by asking them which hand they typically use to complete activities of daily living, such as writing, throwing a ball, cutting paper with scissors, brushing teeth, and eating with a spoon. Participants can answer if they would use strictly their right hand, right more than left, both equally, left more than right, or strictly their left hand. Participants are then categorized as left-handed, ambidextrous, or right-handed.
Action Research Arm Test (ARAT) | Assessment occurs at one cross-sectional timepoint within 2 weeks of research consent
  This test is used to assess upper limb performance post-stroke by measuring coordination, dexterity, and functioning. Participants are asked to complete tasks grouped into four categories - gross movement, grasp, grip, and pinch. Task performance is rated on a four point scale, in which 0 represents no movement and 3 represents normal movement. The Action Research Arm Test has demonstrated an inter-rater reliability between 0.996-0.998.
Modified Ashworth Scale | Assessment occurs at one cross-sectional timepoint within 2 weeks of research consent
  This test is used to assess spasticity at different joints of the upper extremity. The test will be performed at the shoulder, elbow, forearm, wrist, and digits. The six point scale will indicate presence of the abnormal increase in muscle tone, ranging from 0 = no increase in tone to 4 = affected part in rigid flexion and extension. Higher scores on this assessment mean worse outcomes.
Nottingham Sensory Assessment (Erasmus MC) | Assessment occurs at one cross-sectional timepoint within 2 weeks of research consent
  This test is used to understand sensory deficits of the upper extremity. Participants are exposed to distinct stimuli and asked to describe if the object is sharp or blunt and the location of the stimulus. A rater will determine if the reported sensation was absent, impaired, or normal.
National Institute of Health Stroke Scale | Assessment occurs at one cross-sectional timepoint within 2 weeks of research consent
  This test provides information about overall stroke severity. The test includes a series of different questions which allow for the assessment of level of consciousness, vision, facial, arm, and leg motor weakness, sensation, coordination, and language expression and reception. Score range from 0 to 42. Higher scores on this assessment mean worse outcomes.
Montreal Cognitive Assessment (MoCA) | Assessment occurs at one cross-sectional timepoint within 2 weeks of research consent
  This test is used to assess cognitive dysfunction by testing multiple different cognitive domains including attention and concentration, executive functions, memory, language, visuospatial skills, conceptual thinking, calculations, and orientation. Scores range from 0 to 30 with higher scores meaning better cognitive outcome.
Patient Health Questionnaire 9 (PHQ-9) | Assessment occurs at one cross-sectional timepoint within 2 weeks of research consent
  This questionnaire is used to screen, diagnose, and monitor post stroke depression. The questionnaire includes a series of questions which allow a participant to self-report how often he/she has been experiencing symptoms of depression. Scores range from 0 to 27 with higher scores meaning worse depression.
History of TBI | Assessment occurs at one cross-sectional timepoint within 2 weeks of research consent
  This questionnaire is used to collect information about the participant's injury history to his/her head. Participants are asked how many head injuries they have sustained, if any of these events led to loss of consciousness, and a description of their worst head injury.
Barthel Index | Assessment occurs at one cross-sectional timepoint within 2 weeks of research consent
  This test provides information about the participant's level of independence in performing activities of daily living (ADLs). The test includes a series of questions which can be asked of the participant or a caregiver. Scores range from 0 to 100 with higher scores meaning better outcome.
Modified Rankin Scale | Assessment occurs at one cross-sectional timepoint within 2 weeks of research consent
  This scale is used to measure the degree of disability based on functional status. The scale involves a series of questions asked to determine the degree of disability a participant is experiencing at the current timepoint. Scores range from 0 to 6 with higher scores meaning worse outcome.
Defense and Veterans Pain Rating Scale | Assessment occurs at one cross-sectional timepoint within 2 weeks of research consent
  This scale is used to measure a participant's impression of the pain he/she is feeling at the time of assessment. The participant is asked to rate the pain on a scale of 0 to 10, with 0 indicating no pain and 10 being "as bad as it could be".
Manual Muscle Testing | Assessment occurs at one cross-sectional timepoint within 2 weeks of research consent
  This assessment is used to measure the strength of the participant's muscles in his/her upper extremities. Participants are asked to maximally contract these muscles and the force produced is recorded by a dynamometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Providence VA Medical Center, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No